CLINICAL TRIAL: NCT02907567
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Study of the Safety & Pharmacokinetics of Two Doses of CT1812 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Clinical Trial of CT1812 in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG0102
Record Dates: First submitted 2016-09-05; First posted 2016-09-20 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Treatment-Low (Active Comparator): 6 subjects randomized to 280 mg (Low) CT1812
  Interventions: Drug: CT1812
- Active Treatment-High (Active Comparator): 6 subjects randomized to 560 mg (High) CT1812
  Interventions: Drug: CT1812
- Placebo (Placebo Comparator): 4 subjects randomized to matching placebo of CT1812
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT1812 — Active study drug
  Other Names: Study Drug
  Arms: Active Treatment-High; Active Treatment-Low
Drug: Placebo — non-active study drug
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel group study of two doses of CT1812 in adults with mild to moderate Alzheimer's Disease to evaluate the safety and tolerability of oral CT1812, administered for 28 days. This trial may include up to 8 qualified investigator sites in Australia.

DETAILED DESCRIPTION:
Screening procedures will occur up to 42 days. Eligible subjects will randomized at the clinic on Day 1 and receive the first dose of study drug. Dosing for 28 days thereafter off-site and a total of 5 clinic visits over the treatment period for safety and lab assessments. Then a 7 day post-treatment completion follow-up visit (Day 35) and End of Study for last safety assessments (Day 49).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to initiation of any study-related procedures. For subjects unable to provide written consent, consent will be provided by the Person Responsible per local regulations.
2. Men and women, 50-80 years in age inclusively with a diagnosis of mild to moderate Alzheimer's disease according to the 2011 NIA-AA. Women must be neither pregnant nor nursing, and are either surgically sterile, postmenopausal or premenopausal using an acceptable method of contraception.
3. Previous decline in cognition for more than six months.
4. Neuroimaging (MRI) obtained within the previous 6 months or during screening, consistent with the clinical diagnosis of Alzheimer's disease.
5. MMSE 18-26 inclusive.
6. No active depression and a Geriatric Depression Score (GDS) of < 6.
7. Modified Hachinski Ischemia score ≤ 4.
8. Formal education of eight or more years.
9. Living at home or in a community setting (assisted living) without continuous nursing care. Each subject must have a reliable caregiver who sees them at least 3 times weekly, can oversee the administration of study drug, and is willing and able to participate in all clinic visits and some study procedures. Responsible caregiver must provide written informed consent to participate.
10. Concurrent use of acetylcholinesterase inhibitors or memantine must be stable for 90 days prior to screening and not expected to change.

Exclusion Criteria:

1. History of or screening brain MRI scan indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor such as meningioma).
2. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia,
   2. Other neurodegenerative condition
   3. Seizure disorder
   4. Other infectious, metabolic or systemic diseases affecting the central nervous system
3. A current DSM-V diagnosis of active major depression, schizophrenia or bipolar disorder.
4. Clinically significant, advanced or unstable disease that may interfere with outcome measures, and which may bias the assessment of the clinical or mental status of the patient or put the patient at special risk

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Incidence and review of Treatment Emergent Adverse Events | Up to 30 days
  Treatment Emergent Adverse Events will be assessed by reviewing: Physical Exams; monitoring of vital signs, ECGs, and clinical and laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Michael Woodward, MD, Principal Investigator — Austin Health
Locations (4):
- Australia (4):
  - Dr. Phillip Morris, Southport, Queensland
  - Austin Health, Ivanhoe, Victoria
  - Epworth Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital Hospital, Parkville, Victoria

REFERENCES:
- [Derived] Izzo NJ, Yuede CM, LaBarbera KM, Limegrover CS, Rehak C, Yurko R, Waybright L, Look G, Rishton G, Safferstein H, Hamby ME, Williams C, Sadlek K, Edwards HM, Davis CS, Grundman M, Schneider LS, DeKosky ST, Chelsky D, Pike I, Henstridge C, Blennow K, Zetterberg H, LeVine H 3rd, Spires-Jones TL, Cirrito JR, Catalano SM. Preclinical and clinical biomarker studies of CT1812: A novel approach to Alzheimer's disease modification. Alzheimers Dement. 2021 Aug;17(8):1365-1382. doi: 10.1002/alz.12302. Epub 2021 Feb 8. PMID 33559354